CLINICAL TRIAL: NCT04203420
Title: Prevalence of Primary Aldosteronism in Young Adults With Acute Stroke
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Head of Department of Endocrinology, Chongqing Medical University
Other Study IDs: PASTROKE
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with PA: patients who finally been diagnosed with primary aldosteronism
  Interventions: Other: screening and confirmatory tests
- patients without PA: patients who finally been diagnosed without primary aldosteronism
  Interventions: Other: screening and confirmatory tests

INTERVENTIONS:
Other: screening and confirmatory tests — screening test is a blood test of the ratio of plasma aldosterone concentration(PAC) and direct renin concentration(DRC), confirmatory test is Captopril Challenge test

SUMMARY:
The guideline requires clinical works to screen for primary aldosteronism(PA) in young adults with family history of stroke at early onset. But the prevalence of PA in young adults with stroke onset before 45 years old had never been investigated. The study aimed to discover the prevalence as well as the clinical characteristics between patients with PA and those without PA during stroke attack. In order to fulfill this objective, investigators intended to conduct a cross-sectional study by taking screening and confirmatory tests among young adults who once admitted due to early onset of acute stroke.

ELIGIBILITY:
Inclusion Criteria:

- patients who were once admitted in the First affiliated hospital of Chongqing Medical university(CQMU), with stroke onset less than two weeks

Exclusion Criteria:

death, serious sequela with motor, comprehensive or linguistic dysfunction, patients unwilling to join in, etiology of trauma, infective or tumor disease, patients with impaired cardiac, renal or liver function during admission-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who were once admitted in the First affiliated hospital of CQMU during Jan.2006 to Feb.2019 with stroke onset less than two weeks. Age between 18 to 45y.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
prevalence of PA | through study completion, an average of 2 years
  to find out the proportion of PA patients in young adults with early onset of acute stroke

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided